CLINICAL TRIAL: NCT00402935
Title: Effects of Cytotoxic Chemotherapy on Ovarian Structure and Function
Brief Title: Ovarian Damage in Young Premenopausal Women Undergoing Chemotherapy for Cancer
Status: Withdrawn | Type: Observational
Why Stopped: slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marjorie Greenfield, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CWRU3803; P30CA043703 (NIH); CASE-CWRU-3803 (Other: Case Comprehensive Cancer Center); CASE-01-04-15
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Leukemia; Long-term Effects Secondary to Cancer Therapy in Adults; Long-term Effects Secondary to Cancer Therapy in Children; Lymphoma; Sexual Dysfunction and Infertility; Sexuality and Reproductive Issues; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: long-term effects secondary to cancer therapy in adults; long-term effects secondary to cancer therapy in children; sexual dysfunction and infertility; sexuality and reproductive issues; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; secondary acute myeloid leukemia; stage I adult Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; childhood acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Lymphoma; Sexual Dysfunction, Physiological; Infertility; Sexuality; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Hodgkin Disease; Recurrence; Congenital Abnormalities | interventions — Therapeutics; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection at the same time points for follicle-stimulating hormone, estradiol, and inhibin B levels.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: laboratory biomarker analysis — Patients undergo blood collection at the same time points for follicle-stimulating hormone, estradiol, and inhibin B levels.
Procedure: fertility assessment and management — Patients undergo a transvaginal or transabdominal ultrasound to measure the ovarian volume and count the number of antral follicles.
Procedure: management of therapy complications — Patients are also asked to fill out questionnaires on estrogen-depletion symptoms at those times. Patients also keep a calendar of menstrual bleeding and hormonal medications.
Procedure: ultrasound imaging — Patients undergo a transvaginal or transabdominal ultrasound to measure the ovarian volume and count the number of antral follicles.

SUMMARY:
RATIONALE: Comparing results of diagnostic procedures, such as ultrasound, done before, during, and after chemotherapy may help doctors learn about the side effects of chemotherapy and help plan the best treatment.

PURPOSE: This clinical trial is studying ovarian damage in young premenopausal women undergoing chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence and timing of ovarian dysfunction/damage in younger premenopausal women undergoing cytotoxic chemotherapy for cancer.
* Determine the feasibility of a prospective, randomized study to assess if gonadotropin analogues can protect the ovary from the cytotoxic effects of chemotherapy.
* Determine the number of patients required for adequate power to test the hypothesis.

OUTLINE: This is a pilot, prospective study.

Patients undergo a transvaginal or transabdominal ultrasound to measure the ovarian volume and count the number of antral follicles at baseline, 3 months after beginning cytotoxic chemotherapy, and at 6 months after completion of treatment. Patients undergo blood collection at the same time points for follicle-stimulating hormone, estradiol, and inhibin B levels. Patients are also asked to fill out questionnaires on estrogen-depletion symptoms at those times. Patients also keep a calendar of menstrual bleeding and hormonal medications.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer, including, but not limited to, any of the following:

  * Acute lymphocytic leukemia
  * Acute myeloid leukemia
  * Hodgkin's lymphoma
* Must have primary disease with significant chance for long-term survival after therapy
* Scheduled to receive chemotherapeutic agents known to be associated with ovarian failure, including any of the following:

  * Cyclophosphamide
  * Mechlorethamine hydrochloride
  * Busulfan
  * Procarbazine hydrochloride
  * Chlorambucil
  * Melphalan
  * Ifosfamide
  * Cisplatin
  * Carboplatin
* Postmenarchal and premenopausal

PATIENT CHARACTERISTICS:

* Female
* Weight ≤ 250 pounds
* Not pregnant

PRIOR CONCURRENT THERAPY:

* No prior or concurrent total-body irradiation or radiotherapy to the pelvis
* Concurrent bone marrow transplantation allowed
* Concurrent oral contraception and/or gonadotropin releasing-hormone analogue allowed

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: premenopausal women undergoing chemotherapy for cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Incidence of ovarian damage after cytotoxic chemotherapy as determined by changes in ovarian volume, antral follicle count, and follicle-stimulating hormone, estradiol, and inhibin B levels | Ultrasound to measure the ovarian volume and count the number of antral follicles at baseline, 3 months after beginning cytotoxic chemotherapy, and at 6 months after completion of treatment. Patients undergo blood collection at the same time points.

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Greenfield, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00402935?term=cwru3803&rank=1